CLINICAL TRIAL: NCT04765449
Title: Third-Party COVID-19-Specific Cytotoxic T Lymphocytes for the Treatment of Elderly and High-Risk Patients With COVID-19 Infection
Brief Title: Transfer of Infection Fighting Immune Cells Generated in the Laboratory to High Risk Patients With COVID-19 Infection
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Thomas Jefferson University (Other)
Collaborators: Tevogen Bio Inc (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 21P.015; JT 16697 (Other: JeffTrial Number)
Record Dates: First submitted 2021-02-19; First posted 2021-02-21 (Actual); Last update posted 2025-04-29 (Actual); Status verified 2025-04

CONDITIONS: Covid19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- ARM A: Covid-19 Patients Receiving CTLs (Experimental): Patients who have an HLA antigen in common with COVID-19 fighting T cells will receive the COVID-19 T cells. They will be premedicated with diphenhydramine and acetaminophen before the cells are infused intravenously. Close monitoring will continue in the patients' homes for 14 days. Three to six patients will receive a specific dose of T cells, and then if there are no serious side effects, the dose will be increased for the next group of patients. There are 4 doses of T cells to be tested, and each patient will complete a 14 day monitoring period before the next patient can be treated.
  Interventions: Drug: Cytotoxic T Lymphocytes
- ARM B: Covid-19 Patients Not Receiving CTLs (No Intervention): Patients in the observation arm will not have inherited an HLA antigen in common with the COVID-19 T cells and so cannot receive the T cells. They will be monitored by the study staff for the 14 day monitoring period in their homes. They will be taught to record their own blood pressure, temperature, and oxygen level (pulse oximetry) at home and report this information, as well as their progress in getting over the COVID-19 infection, to the study staff every day by phone. The outcomes of patients on arm B will be compared to the outcomes of patients treated on Arm A to see if the T cells made a difference in how patients recovered from COVID-19. Patients in Arm B are not prevented from being treated with any available COVID-19 therapy.

INTERVENTIONS:
Drug: Cytotoxic T Lymphocytes — Given IV. Cytotoxic T Lymphocytes collected from healthy volunteer donors who have recovered from COVID-19. The T cells are collected, manufactured to be COVID-specific, and stored frozen at Thomas Jefferson University.
  Other Names: CTLs
  Arms: ARM A: Covid-19 Patients Receiving CTLs

SUMMARY:
This clinical trial will study the safety and efficacy of COVID-19-specific T cells when given as treatment to adult patients (age ≥ 18 years) with a COVID-19 infection. This immunologic treatment is aimed at patients, who are at high risk of progression due to their advanced age, or other underlying health conditions. The outcomes of patients receiving the T cells (Arm A) will be compared to patients treated with standard of care (Arm B).

DETAILED DESCRIPTION:
T cells that recognize COVID-19 peptides will be manufactured at Thomas Jefferson University and are frozen and ready for use. The T cells have to have an immune protein called HLA in common with a patient to work. If a patient enrolled on the COVID-19 study has this HLA, they will receive a dose of the COVID-19 T cells. Groups of 3-6 patients will be treated at each testing dose level. There are four dose levels of T cells: 1 x 105/kg, 3 x 105/kg, 1 x 106/kg, and 3 x 106/kg. Patients will receive the T cells intravenously in the hospital and be monitored there for 4 days before being discharged. Before discharge, patients will be taught to take and record their temperature, blood pressure, and oxygen levels (using a finger monitor) at home. After discharge, study staff will continue to monitor patient symptoms and recordings with video visits or phone calls daily until the monitoring period of 14 days is over. Patients will also be asked to give blood samples 7, 14, 28, days and 2, 3, and 6 months after the T cells are given. Patients who meet study criteria and wish to participate but do not have the HLA protein in common with the T cells, will be monitored by study personnel in their own homes for the full 14 day period. These patients will also be taught to take and record their temperature, blood pressure, and oxygen level. Study personnel will contact them daily by video or voice calls and check on the results of their readings and their symptoms. These patients may be treated with any standard or experimental COVID-19 therapy. How patients handle their COVID-19 infection will be compared between the group of people receiving the T cells and the group of people who do not receive the T cells.

ELIGIBILITY:
Inclusion Criteria:

Have a documented active COVID-19 infection and one of the following high-risk criteria:

* Malignancy receiving radiation or chemotherapy in the prior 24 months.
* Chronic lung disease such as asthma, COPD, interstitial lung disease, pulmonary hypertension or cystic fibrosis, requiring treatment beyond inhaled medications
* Hypertension either treated or with evidence of need for treatment
* Cardiovascular disease requiring active medical monitoring and care including heart failure, heart dysrhythmias, coronary artery disease, congenital heart disease, cardiomyopathy, or pulmonary hypertension
* History of ischemic stroke
* Diabetes (type 1, type 2, or gestational) requiring treatment with insulin or oral hypoglycemics
* Chronic Kidney Disease (Hx of stage 3b or greater as defined by the National Kidney Foundation)
* Chronic Liver Disease (Previously diagnosed with cirrhosis or previously classified as having Pugh-Child class A-C liver disease) oObesity (BMI >= 35) oSickle Cell Disease or Thalassemia
* Patients requiring nursing home support or who have a Karnofsky Performance Status of 70% or less antedating their COVID-19 illness.
* Age >= 65 (with or without previously identified comorbid conditions)

Exclusion Criteria:

* Matching their intended CTL product donor at 5 or 6 of 6 HLA-class I (HLA-A, B, and C) alleles.
* Requiring supplemental oxygen
* Evidence of active COVID-19-related CRS as evidenced by 2 or more of the following characteristics of cytokine storm:

  o> grade 1 CRS on ASTCT criteria. ASTCT criteria do not provide quantitative guidelines regarding the definition of hypotension. For this trial, hypotension will be defined as:
  1. requiring vasopressors
  2. Systolic blood pressure <90 mm Hg
  3. Diastolic B/P < 60 mm Hg NB Lower systolic and diastolic blood pressures will be acceptable if patient's blood pressure is at his/her known baseline.

     * Uncontrolled hypertension as defined by a systolic pressure of > 180 mm Hg or diastolic pressure > 100 mm Hg. A second blood pressure reading may be obtained by study personnel to assure blood pressure accuracy.
     * radiographic studies consistent with adult respiratory distress syndrome
     * Patients requiring acute dialysis
     * hyperferritinemia as defined by ferritin > 2000 ng/mL 55
     * Concurrent treatment with >5 mg of prednisone daily (or equivalent).
* Current or ongoing administration of calcineurin inhibitors, chemotherapy, radiation, or other immunosuppressive agents.

  * That cannot be held for 14 days after CTL infusion
  * That would not decay 3 1/2 half-lives by the day of CTL infusion using longest published half-life.
* Receipt of agents with ongoing immunosuppressive properties in the last 30 days including, ATG, Alemtuzumab, or similar agents.
* Prior allogeneic bone marrow, stem cell, or solid organ transplant. Patients with a history of autologous transplant are eligible for study if one year has elapsed since their transplant.
* Active HIV infection with CD4 count less than 200/ul.
* Pregnancy (lactating females allowable)
* Concomitant treatment with another experimental intervention for COVID-19 other than Remdesivir.
* History of allergic reaction to cellular therapy products (includes blood transfusion), diphenhydramine, or tocilizumb
* Corrected QT interval > 450 milliseconds
* History of torsade de pointes or other ventricular arrhythmia Women of childbearing potential, and partners of women of childbearing potential should be using at least one method of highly effective contraception at the time of enrollment and for the 14-day duration of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2021-09-15 (Actual); Primary Completion 2022-07-29 (Actual); Study Completion 2023-01-19 (Actual)

PRIMARY OUTCOMES:
Safety of COVID-19-specific CTLs: Infusion Reactions | Within 48 Hours of CTL Infusion
  Safety will be measured by the absence of: Grade ≥ 3 acute infusion reactions
Safety of COVID-19-specific CTLs: Grade 4 AEs | Within 14 days of CTL infusion
  Safety will be measured by the absence of: Any grade 4 or higher adverse event thought to be related to the CTL therapy and outside the spectrum of identified COVID related events.
Safety of COVID-19-specific CTLs: GVHD | Within 14 days of CTL infusion
  Safety will be measured by the absence of: Any manifestation of acute GVHD (for acute grades 2-4 GVHD-Glucksberg criteria) 53 resistant to 2 mg/kg of solumedrol or equivalent
Safety of COVID-19-specific CTLs: Marrow Aplasia | Within 14 days of CTL infusion
  Safety will be measured by the absence of: Marrow aplasia due to 3rd party engraftment
Safety of COVID-19-specific CTLs: Neurotoxicty | Within 14 days of CTL infusion
  Safety will be measured by the absence of: Grade ≥ 2+ Neurotoxicity as measured by the ASTCT/ICANS consensus grading system
Safety of COVID-19-specific CTLs: CRS | Within 14 days of CTL infusion
  Safety will be measured by the absence of: Grade ≥ 2+ CRS as measured by the ASTCT Consensus Grading Criteria for CRS

SECONDARY OUTCOMES:
Measurement of COVID-19 viral load | Up to 14 Days
  Patients will have blood drawn, nasal (not nasopharyngeal) specimens collected
Studies to detect the persistence of the COVID-19-specific T cells after COVID-19 T cell infusion | Up to 6 months
  Patients will have blood drawn, nasal (not nasopharyngeal) specimens collected
Studies to examine the development of endogenous COVID-19 specific T cells | Up to 6 months
  Patients will have blood drawn, nasal (not nasopharyngeal) specimens collected
Studies to examine the development of anti-COVID-19 antibodies | Up to 6 months
  Patients will have blood drawn, nasal (not nasopharyngeal) specimens collected
Review of medical history including the need for supplemental oxygen, the ability to return to work, performance status, grade of dyspnea, grade of fatigue, survival, the need for blood pressure support | Up to 6 months
  Patients will have their medical course followed by the study team

CONTACTS AND LOCATIONS:
Locations (1):
- Thomas Jefferson University, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Grosso D, Wagner JL, O'Connor A, Keck K, Huang Y, Wang ZX, Mehler H, Leiby B, Flomenberg P, Gergis U, Nikbakht N, Morris M, Karp J, Peedin A, Flomenberg N. Safety and feasibility of third-party cytotoxic T lymphocytes for high-risk patients with COVID-19. Blood Adv. 2024 Aug 13;8(15):4113-4124. doi: 10.1182/bloodadvances.2024013344. PMID 38885482